CLINICAL TRIAL: NCT01973270
Title: Community-Based Cognitive Training in Early Schizophrenia
Acronym: COTES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH102063-01 (NIH)
Record Dates: First submitted 2013-08-06; First posted 2013-10-31 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Targeted Cognitive Training - TCT (Experimental): Neuroadaptive cognitive training
  Interventions: Behavioral: Neuroadaptive cognitive training
- General Cognitive Exercises (GCE) (Experimental): Neuroadaptive cognitive training
  Interventions: Behavioral: Neuroadaptive cognitive training
- Treatment as Usual (No Intervention): Treatment as Usual

INTERVENTIONS:
Behavioral: Neuroadaptive cognitive training — TCT exercises consist of three modules: an Auditory Processing Module (40-50 hours of training); a Visual Processing Module (30 hours); a Cognitive Control Module prototype (20 hours). [Based on the results of our current RCT, Posit Science has revised aspects of the training modules in order to further optimize its effectiveness for treatment of schizophrenia. In this study, we will use updated versions of the training software: an Auditory Module (20 hours), and a Social Module (10 hours). Features from the Cognitive Control module prototype have been expanded and incorporated into these new modules.
  Arms: General Cognitive Exercises (GCE); Targeted Cognitive Training - TCT

SUMMARY:
The purpose of this study is to determine whether cognitive training exercises can improve cognitive functioning in young patients with recent-onset schizophrenia, schizoaffective, schizophreniform, and psychosis NOS who are being treated in community mental health settings. We will investigate the effects of web-based cognitive training exercises delivered on a portable laptop computer. The findings will provide us with valuable information on whether cognitive training can improve the cognition and functioning of young individuals early in the course of schizophrenia.

DETAILED DESCRIPTION:
The purpose of this study is to perform a double-blind randomized controlled trial (RCT) in young patients with recent-onset (RO) schizophrenia to target improvement in cognitive functioning within real-world treatment settings. This multi-site study will be performed in 4 community mental health centers with specialized Early Intervention Services (EIS). We will compare the effects of web-based targeted cognitive training (TCT) vs. web-based general cognitive exercises (GCE), both delivered via portable laptop computers. We will investigate the behavioral and functional changes seen immediately after the intervention as well as at 6-month follow-up, compared to a no-training control group (NTC). This will be the first study to investigate cognitive enhancement for young RO schizophrenia patients in community mental health settings, using scalable interactive neurotechnology, and the first to compare two distinct cognitive training approaches. This study will generate high impact data on the potential for targeted pre-emotion of the downward spiral of in cognitive and functional disability that often characterizes psychotic illness. It will also generate valuable data on the relative effects of two distinct cognitive training approaches in schizophrenia, each derived from a very different theoretical rationale, providing much-needed information on the efficacy of a targeted "distributed neural system" training model derived from systems neuroscience vs. a "general cognitive stimulation" training model derived from neuropsychological rehabilitation approaches.

The aims of this project are based on the current state of early psychosis research, as well as our own experience successfully applying neuroscience-informed cognitive training in schizophrenia. It is now abundantly clear that cognitive/neural system dysfunction represents a significant risk factor for schizophrenia as well as a poor prognostic indicator. Functional outcome in RO schizophrenia is predicted by level of cognitive impairment and baseline cognitive reserve, and recent findings suggest that specialized EIS programs focusing only on symptom reduction and psychosocial support may not robustly improve long-term outcomes- indicating that critical treatment targets are not being addressed at present in early psychosis interventions. Cognitive dysfunction and underlying neural system inefficiency should therefore be one of the primary targets for pre-emptive intervention in early psychosis. In this study, we will determine whether we can achieve this goal using cognitive training delivered via a portable computer, in order to improve functional outcome in young individuals with RO schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia, schizoaffective disorder, psychosis Not Otherwise Specified (NOS), Unspecified Schizophrenia Spectrum Disorder, Schizophrenia Spectrum Disorder, Specified, or schizophreniform disorder with onset of first psychotic episode within the last 2 years.
* Good general physical health
* Between 18 and 35 years of age
* Is fluent and proficient in the English language
* Currently enrolled in PREP/BEAM services
* Achieved clinical stability (e.g., outpatient status for at least 1 month before study entry)

Exclusion Criteria:

* Any neurological disorder
* If clinically significant substance abuse occurs that is impeding the subject's ability to participate fully during recruitment, assessment, or training, the subject will be dropped from the study.
* Being treated with benztropine, diphenhydramine, or high doses of clozapine (>500 mg po qd) or olanzapine(to be determined on a case by case basis)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2013-12; Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Neurocognition | Baseline, Post-Training, 6 month Follow-up
  Neurocognition will be assessed using the MATRICS Consensus Cognitive Battery [MCCB]. The MCCB assesses the following domains of neurocognitive functioning: 1) Speed of Processing, 2) Attention/Vigilance, 3) Working Memory, 4) Verbal Learning, 5) Visual Learning, 6) Reasoning and Problem Solving; and 7) Social Cognition. We will also assess Verbal Memory (HVLT delayed recall), Visual Memory (BVMT delayed recall), and administer an additional measure of Reasoning and Problem Solving [BACS Tower of London]. In addition to the MCCB measure of social cognition, we will assess the following constructs: affect recognition, emotional prosody [Penn Prosody Identification, and theory of mind [Faux Pas test.7 hours spread over 3 appointments in a 1-2 week period, 5 hours post-training and an additional 5 hours at a 6-month follow-up.
Functioning | Baseline, Post-Training, 6 Month Follow-up
  The Quality of Life Scale-Abbreviated will be our primary outcome measure of functional status. This measure assesses quality of life using subjective questions regarding life satisfaction and objective indicators of social and occupational functioning.
Auditory Processing Speed | Baseline, 10 hours of training
  Early target engagement is the degree to which an individual demonstrates initial performance improvement ("learning") upon exposure to training. Early target engagement will be measured by auditory processing speed during cognitive training exercises.
Reward Sensitivity | Baseline
  The Temporal Experience of Pleasure Scale (TEPS) will be used to assess reward sensitivity.

SECONDARY OUTCOMES:
Functional Capacity | Baseline, Post-Training, 6 Month Follow-up
  Secondary measures of functional capacity/status will include the following MATRICS-recommended measure: The UCSD Performance Based Skills Assessment [UPSA-Brief].
Social Functioning | Baseline, Post-Training, 6 Month Follow-up
  Secondary measures of social functioning will include: The Social Functioning Scale.
Internalized Stigma | Baseline, Post-Training, 6 Month Follow-up
  In order to measure internalized stigma, a component of recovery, we will use the Internalized Stigma of Mental Illness (ISMI) Scale.

OTHER OUTCOMES:
Feasibility and Acceptability | Post-Training (6 weeks)
  We will measure and compare the feasibility and acceptability of the cognitive training programs integrated in the EIS through 1) attrition rates; 2) time to completion of training; 3) user and clinician ratings of acceptability. At post-training (6 weeks), subjects will complete a Likert-type questionnaire composed of elements of a measure used previously by Brain Plasticity Institute to evaluate acceptability for their cognitive training software, and components of a measure we have used previously to assess acceptability of training in our recent-onset RCT. Items assess user experience and satisfaction with the programs, the web-based administration, and the training schedule. Clinicians and family members will complete a Likert-type questionnaire that assess their experience in supporting the clients to use the program, perceived impact on the clients, and the likelihood of using the program outside of a research study.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Prevention and Recovery in Early Psychosis (PREP) Program, San Francisco, California, United States